# 19-012665

# Pre-analytical Factors Affecting ctDNA Analysis in Early and Locally-advanced Breast Cancer

NCT05945290

Document Date: 09/24/2024



Approval Date: September 24, 2024

# RESEARCH PARTICIPANT CONSENT AND PRIVACY AUTHORIZATION FORM

**Study Title:** Pre-analytical factors affecting ctDNA analysis in early and locally advanced

breast cancer

**IRB#:** 19-012665

Principal Investigator: Dr. Pockaj and Colleagues

#### **Key Study Information**

This section provides a brief summary of the study. It is important for you to understand why the research is being done and what it will involve before you decide. Please take the time to read the entire consent form carefully and talk to a member of the research team before making your decision. You should not sign this form if you have any questions that have not been answered. This is a research study. Being in this research study is your choice; you do not have to participate. If you decide to join, you can still stop It's Your Choice at any time. You should only participate if you want to do so. You will not lose any services, benefits or rights you would normally have if you choose not to take part. The purpose of this study is to collect blood and tissue samples for the research of cancer to evaluate the impact of blood collection/processing and long-term storage. **Research Purpose** You are being asked to take part in this research study because you have breast cancer and will be getting treatment for your cancer. Study participation involves 5 blood samples will be collected: 1. Prior to the initiation of your breast cancer treatment as indicated by your treating physician, 2. After your surgery 3. Completion of chemotherapy What's Involved 4. After Radiation therapy (if applicable), if not at 9 months 5. First routine clinical follow up after completion of treatment which is about 1 year. Your tissue from your diagnostic biopsy and surgery will be retrospectively collected for comparative analysis.



# Approval Date: September 24, 2024

| | You will not be required to undergo additional biopsy or surgical procedures as part of this study. |
|---|---|
| | In addition to the collection of blood and tissue, information from your medical record will be collected and stored in a password-protected electronic database. |
| | You will be in the study for as long as it takes to complete your blood draws for the study. |
| | The risks of drawing blood include pain, bruising, lightheadedness, and/or fainting, or rarely, infection at the site of the needle stick. |
| Key Information | This study involves testing your DNA, which is the genetic information you inherited from your parents (also known as genetic testing). You will not be notified of the genetic test results and they will not be put into your medical record. |
| | There are no costs to you for being in the study. |
| | The goal of the study is to gather information; you will not directly benefit from participation. |
| Learn More | If you are interested in learning more about this study, read the rest of this form carefully. The information in this form will help you decide if you want to participate in this research or not. A member of our research team will talk with you about taking part in this study before you sign this form. If you have questions at any time, please ask us. |

# **Making Your Decision**

Taking part in research is your decision. Take your time to decide. Feel free to discuss the study with your family, friends, and healthcare provider before you make your decision. Taking part in this study is completely voluntary and you do not have to participate.

If you decide to take part in this research study, you will sign this consent form to show that you want to take part. We will give you either a printed or electronic copy of this form to keep.

For purposes of this form, Mayo Clinic refers to Mayo Clinic in Arizona, Florida and Rochester, Minnesota; Mayo Clinic Health System; and all owned and affiliated clinics, hospitals, and entities.



Approval Date: September 24, 2024

Name and Clinic Number

# **Contact Information**

| If you have questions about | You can contact |
|---|---|
| <ul> <li>Study tests and procedures</li> <li>Materials you receive</li> <li>Research-related appointments</li> </ul> | Principal Investigator: Barbara Pockaj, M.D. Phone: (480) 301-8000 |
| Research-related concern or complaint | Study Team Contact: Shanann Avelar |
| <ul><li>Research-related injuries or emergencies</li><li>Withdrawing from the research study</li></ul> | <b>Phone:</b> (480) 301-8000 |
| - | Institution Name and Address: |
| | Mayo Clinic |
| | 5777 E Mayo Boulevard |
| | Phoenix, AZ 85054 |
| ■ Rights of a research participant | Mayo Clinic Institutional Review Board (IRB) Phone: (507) 266-4000 |
| | Toll-Free: (866) 273-4681 |
| <ul><li>Rights of a research participant</li></ul> | Research Subject Advocate (RSA) |
| <ul> <li>Any research-related concern or complaint</li> </ul> | (The RSA is independent of the Study Team) |
| <ul> <li>Use of your Protected Health Information</li> </ul> | <b>Phone:</b> (507) 266-9372 |
| <ul> <li>Stopping your authorization to use your<br/>Protected Health Information</li> </ul> | <b>Toll-Free:</b> (866) 273-4681 |
| <ul> <li>Withdrawing from the research study</li> </ul> | E-mail: researchsubjectadvocate@mayo.edu |
| <ul><li>Billing or insurance related to this research<br/>study</li></ul> | Patient Account Services |
| • | <b>Toll-Free:</b> (844) 217-9591 |



**Approval Date:** September 24, 2024

## Why are you being asked to take part in this research study?

You are being asked to take part in this research study because you have breast cancer and will be getting treatment for your cancer.

The plan is to have about 120 people take part in this study at Mayo Clinic.

#### Why is this research study being done?

The purpose of this study is to collect blood and leftover tissue samples for the research of cancer to evaluate the impact of blood collection/processing and long-term storage.

#### Information you should know

#### Who is Funding the Study?

National Institutes of Health and Mayo Clinic are funding the study. National Institutes of Health and Mayo Clinic will pay the institution to cover costs related to running the study.

### How long will you be in this research study?

You will be in the study for as long as it takes to complete your blood draws for the study.

#### What will happen to you while you are in this research study?

If you agree to be in the study, you will be asked to participate in the following: Study participation involves blood samples (approximately 8 tablespoons total) to be collected over the course of about one year at 5 time points depending on your standard of care therapy. If you undergo neoadjuvant therapy, additional blood (approximately 1 ½ tablespoons) will be collected prior to your treatment. The five time points are:



#### Approval Date: September 24, 2024

- 1. Prior to the initiation of your breast cancer treatment as indicated by your treating physician,
- 2. After your surgery
- 3. Completion of chemotherapy
- 4. After Radiation therapy (if applicable), if not at 9 months
- 5. First routine clinical follow up after completion of treatment which is about 1 year.

You will also have routine tests as part of care which will include imaging (mammograms, CT scans) and other blood tests prior to starting treatment. Information will be obtained from your medical record for this research.

Your tissue from your diagnostic biopsy and surgery will be retrospectively collected for comparative analysis. You will not be required to undergo additional biopsy or surgical procedures as part of this study

Tests done only for research purposes are not meant to provide clinical information or help care for you. The results are only important for research. Therefore, the results of tests done with your information and samples will not be provided to you. In the rare event that a finding might affect the health of you or your family, we will contact you and you can choose whether to receive or refuse the information. If you decide to follow up and further medical testing or care is needed, the costs will be billed to you or your insurance.

#### What are the possible risks or discomforts from being in this research study?

The risks of drawing blood include pain, bruising, lightheadedness, and/or fainting, or rarely, infection at the site of the needle stick.

As with all research, there is a chance that confidentiality could be compromised; however, we take precautions to minimize this risk.

Your doctor will discuss the risks of mammograms, CT scans (imaging) as these tests and procedures are part of your standard clinical care.

This study involves testing your DNA, which is the genetic information you inherited from your parents (also known as genetic testing). This testing may include whole genome sequencing (mapping your entire genetic code). You will not be notified of the genetic test results and they will not be put into your medical record.



**Approval Date:** September 24, 2024

A Federal law, called the Genetic Information Nondiscrimination Act (GINA), generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. This law generally will protect you in the following ways:

- Health insurance companies and group health plans may not request your genetic information that we get from this research.
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums.
- Employers with 15 or more employees may not use your genetic information when making a decision to hire, promote, or fire you or when setting the terms of your employment.

All health insurance companies and group health plans must follow this law.

Be aware that this new Federal law doesn't protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance.

#### Are there reasons you might leave this research study early?

You may decide to stop at any time. You should tell the Principal Investigator if you decide to stop and you will be advised whether any additional tests may need to be done for your safety. In addition, the Principal Investigator or Mayo Clinic may stop you from taking part in this study at any time:

- If it is in your best interest,
- If you don't follow the study procedures,
- If the study is stopped.

If you leave this research study early, or are withdrawn from the study, no more information about you will be collected; however, information already collected about you in the study may continue to be used.

We will tell you about any new information that may affect your willingness to stay in the research study.



Approval Date: September 24, 2024

## What if you are injured from your participation in this research study?

#### Where to get help:

If you think you have suffered a research-related injury, you should promptly notify the Principal Investigator listed in the Contact Information at the beginning of this form. Mayo Clinic will offer care for research-related injuries, including first aid, emergency treatment and follow-up care as needed.

#### Who will pay for the treatment of research related injuries:

Care for such research-related injuries will be billed in the ordinary manner, to you or your insurance. Treatment costs for research-related injuries not covered by your insurance will be paid by Mayo Clinic.

## What are the possible benefits from being in this research study?

You won't benefit from taking part in this research study. It is for the benefit of research.

# What alternative do you have if you choose not to participate in this research study?

This study is only being done to gather information. You may choose not to take part in this study.

# What tests or procedures will you need to pay for if you take part in this research study?

You won't need to pay for tests and procedures which are done just for this research study. These tests and procedures are:

• Blood Draws for research



**Approval Date:** September 24, 2024

However, you and/or your insurance will need to pay for all other tests and procedures that you would have as part of your clinical care, including co-payments and deductibles. These tests and procedures are:

- Withdrawal of tissue and blood samples which are clinically indicated for diagnostic purposes.
- Imaging (MRI and CT scan)

You will also be responsible for any co-payments and deductibles.

If you have billing or insurance questions call Patient Account Services at the telephone number provided in the "Contact Information" section of this form.

#### Will you be paid for taking part in this research study?

You won't be paid for taking part in this study.

There is a very small chance that some commercial value may result from the use of your sample. This could include new products like a drug or a test to diagnose a disease. If that happens, you will not be offered a share in any profits.

#### Will your information or samples be used for future research?

Unless you give your permission below, your information or samples collected for this study will not be used or shared for future research, even if the identifiable information such as your name, Mayo Clinic number or date of birth is removed.

We would like to keep your information and samples for future research. You can still take part in this current study even if you don't want your information or samples used for future research.

Researchers at Mayo Clinic who aren't involved with this study may ask to use your information and/or samples for future research. Researchers at other institutions may also ask for a part of your information and/or samples for future studies. Unless you indicate otherwise, the future research may be on any topic. No direct benefits to you are expected from the future research. Your information and/or samples will only be shared consistent with your consent, and with all applicable laws and regulations.



| N | ama anc | l Clinic N | Jumhar |
|---|---------|------------|--------|

**Approval Date:** September 24, 2024

If you approve release of your information and/or samples by checking 'yes' below, Mayo may send the information and/or samples to researchers who request them, but Mayo will <u>not</u> send your name, address, phone number, social security number, or any other identifying information with the information and/or samples. Your information and/or samples may be sent with a code, and only the researchers for this study at Mayo Clinic would be able to link the code to you.

Some future studies may examine your DNA, the genetic information you inherited from your parents (genetic testing). If there are findings which may be useful for your health care, the researchers may contact Mayo Clinic, so Mayo Clinic can give you the option of learning the results. You would be given general information on the potential risks, benefits, and costs of choosing to learn about the findings.

To support future research, de-identified genetic information may be placed in databases accessible by the internet. Some of the information may be available to anyone using the internet, and some will be released only to approved researchers. Combined study information (including genomic summary results) may be published, but the information will not identify you.

Even though information traditionally used to identify you will not be shared, people may develop ways in the future to allow someone to link your genetic information back to you. For this reason, confidentiality cannot be guaranteed.

It is also possible that reidentified information could be used in discriminating ways, and there could be additional unknown risks. We will make every effort to protect your confidentiality.

1 I permit my information and samples to be stored and used in future research of Breast

#### Please read the following statements and mark your choices:

| 1 | Mayo Clinic:. | on and samples to be stored a | nd used in future research of Breast |
|---|---|---|---|
| Yes | ☐ No | Please initial here: | |
| - | • | on and samples to be stored a vent, or treat any other health | nd used in future research at Mayo problems: |
| Yes | ☐ No | Please initial here: | _Date: |
| 3. I permit institutions | • | to give my information and sa | amples to researchers at other |
| Yes | ☐ No | Please initial here: | _Date: |



Approval Date: September 24, 2024

You may withdraw your consent for future use of your information and/or samples at any time, by writing to the Principal Investigator at the address provided in the "Contact Information" section of this consent form.

Your information and/or samples would be removed from any repository where they are stored, if possible. Information and/or samples already distributed for research use will not be retrieved.

#### How will your privacy and the confidentiality of your records be protected?

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. This means that the researchers cannot release or use information, documents, or samples that may identify you in any action or suit unless you say it is okay. They also cannot provide them as evidence unless you have agreed. This protection includes federal, state, or local civil, criminal, administrative, legislative, or other proceedings. An example would be a court subpoena.

There are some important things that you need to know. The Certificate DOES NOT stop reporting that federal, state or local laws require. Some examples are laws that require reporting of child or elder abuse, some communicable diseases, and threats to harm yourself or others. The Certificate CANNOT BE USED to stop a sponsoring United States federal or state government agency from checking records or evaluating programs. The Certificate DOES NOT stop disclosures required by the federal Food and Drug Administration (FDA). The Certificate also DOES NOT prevent your information from being used for other research if allowed by federal regulations.

Researchers may release information about you when you say it is okay. For example, you may give them permission to release information to insurers, medical providers or any other persons not connected with the research. The Certificate of Confidentiality does not stop you from willingly releasing information about your involvement in this research. It also does not prevent you from having access to your own information.

Mayo Clinic is committed to protecting the confidentiality of information obtained about you in connection with this research study. Your sample will be stored at Mayo or University of Wisconsin-Madison and would be given a code (instead of your name) while it is stored and when it is used in research. This code allows your sample to be used without anyone knowing that it is your sample just by looking at the label. In addition, all data collected is stored in a password-protected database.



**Approval Date:** September 24, 2024

During this research, information about your health will be collected. Under Federal law called the Privacy Rule, health information is private. However, there are exceptions to this rule, and you should know who may be able to see, use and share your health information for research and why they may need to do so.

Information about you and your health cannot be used in this research study without your written permission. If you sign this form, it will provide that permission (or "authorization") to Mayo Clinic.

#### Your health information may be collected from:

- Past, present and future medical records.
- Research procedures, including research office visits, tests, interviews and questionnaires.

#### Your health information will be used and/or given to others to:

- Do the research.
- Report the results.
- See if the research was conducted following the approved study plan, and applicable rules and regulations.

#### Your health information may be used and shared with:

- Mayo Clinic research staff involved in this study.
- Other Mayo Clinic staff involved in your clinical care.
- The sponsor(s) of this study and the people or groups hired by the sponsor(s) to help perform this research.
- The Mayo Clinic Institutional Review Board that oversees the research.
- Federal and State agencies (such as the Food and Drug Administration, the Department of Health and Human Services, the National Institutes of Health and other United States agencies) or government agencies in other countries that oversee or review research.

#### How your information may be shared with others:

While taking part in this study, you will be assigned a code that is unique to you, but does not include information that directly identifies you. This code will be used if your study information is sent outside of Mayo Clinic. The groups or individuals who receive your coded information will use it only for the purposes described in this consent form.

If the results of this study are made public (for example, through scientific meetings, reports or media), information that identifies you will not be used.



**Approval Date:** September 24, 2024

In addition, individuals involved in study oversight and <u>not</u> employed by Mayo Clinic may be allowed to review your health information included in past, present, and future medical and/or research records. This review may be done on-site at Mayo Clinic or remotely (from an off-site location). These records contain information that directly identifies you. However, the individuals will not be allowed to record, print, or copy (using paper, digital, photographic or other methods), or remove your identifying information from Mayo Clinic.

#### Is your health information protected after it has been shared with others?

Mayo Clinic asks anyone who receives your health information from us to protect your privacy; however, once your information is shared outside Mayo Clinic, we cannot promise that it will remain private and it may no longer be protected by the Privacy Rule.

#### Your Rights and Permissions

Participation in this study is completely voluntary. You have the right not to participate at all. Even if you decide to be part of the study now, you may change your mind and stop at any time. You do not have to sign this form, but if you do not, you cannot take part in this research study.

Deciding not to participate or choosing to leave the study will not result in any penalty. Saying 'no' will not harm your relationship with your own doctors or with Mayo Clinic.

If you cancel your permission for Mayo Clinic to use or share your health information, your participation in this study will end and no more information about you will be collected; however, information already collected about you in the study may continue to be used.

You can cancel your permission for Mayo Clinic to use or share your health information at any time by sending a letter to the address below:

Mayo Clinic
Office for Human Research Protection
ATTN: Notice of Revocation of Authorization
201 Building 4-60
200 1st Street SW
Rochester, MN 55905



**Approval Date:** September 24, 2024

Alternatively, you may cancel your permission by emailing the Mayo Clinic Research Subject Advocate at: researchsubjectadvocate@mayo.edu.

Please be sure to include in your letter or email:

- The name of the Principal Investigator,
- The study IRB number and /or study name, and
- Your contact information.

Your permission for Mayo Clinic to use and share your health information lasts forever, unless you cancel it.

There is no expiration or end date related to the Sponsor's use of your health information received from Mayo Clinic as part of this study.

IRB#: 19-012665 00 E-sign AS Page 13 of 14 IRB Doc. Ctrl # 10013.33



**Approval Date:** September 24, 2024

| ripprovar Date. | September 21, 2021 | |
|---|---|---|
| Enrollment and Permission Signatures Your signature documents your permission to take part in this research. | | |
| Signature | | |
| - | ent the research study to the participant. all questions about this research study to t | the best of my ability. |
| Printed Name | Date (mm/dd/yyyy) | Time (hh:mm am/pm) |
| Signature | | |